CLINICAL TRIAL: NCT07069907
Title: The Improvement of Indoor Air and Health Effects After Air Purifier Intervention Among Susceptible Population in Industrial Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: KMUHIRB-SV(II)-20210120
Record Dates: First submitted 2025-06-22; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Asthma (Diagnosis); COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Asthma; Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: a double-blind, randomized, and crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photocatalytic oxidation intervention (Sham Comparator)
  Interventions: Other: Air purfiers with photocatalytic oxidation (PCO)
- photocatalytic oxidation and filters intervention (Active Comparator)
  Interventions: Other: Air purfiers with photocatalytic oxidation (PCO) + filters

INTERVENTIONS:
Other: Air purfiers with photocatalytic oxidation (PCO) — PCO was proved to decompose gaseous pollutants in chamber studies, while there is no study investigate the effects in real-world. We used PCO air purifiers in households for two weeks.
  Arms: photocatalytic oxidation intervention
Other: Air purfiers with photocatalytic oxidation (PCO) + filters — PCO was proved to decompose gaseous pollutants in chamber studies, while there is no study investigate the effects in real-world. We used PCO and filters air purifiers in households for two weeks, to understand the effects comparing with PCO.
  Arms: photocatalytic oxidation and filters intervention

SUMMARY:
Invesitigators conducted a double-blind, randomized, and crossover study to investigate the effects of PCO and PCO + filters interventions on indoor air pollutants in households and health outcomes in susceptible group, such as asthma and COPD patients.

DETAILED DESCRIPTION:
Invesitigators measured indoor air pollutants, including particulate matter, bioaerosols, gaseous pollutants, in households and health outcomes, including lung function, respiratory symptoms, fractional exhaled nitric oxide, blood pressure, biomarkers, urinary heavy metals, and polycyclic aromatic hydrocarbons, in susceptible group, such as asthma and COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* dianosed with asthma/COPD

Exclusion Criteria:

* did not diagonse with asthma /COPD

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Indoor air pollutants | One day 0 (before intervention) and day 1 (after intervention)
  The DustTrak DRX mass monitor (Model 8533, TSI, Shoreview, MN, USA) was used to measure PM1, PM2.5, PM4, PM10, and TSP continuously for 24 h, and UFPs were measured for 15 min at a time by using the P-Trak Ultrafine Particle Counter (Model 8525, TSI, Shoreview, MN, USA). The YesAir 15-channel indoor air quality monitor (Critical Environment Technologies Canada, Delta, British Columbia, Canada) was used to measure TVOC, NO2, SO2, CO, and CO2 continuously for 24 h.
  Airborne bacteria and fungi were collected using MAS-100 air sampler, which is a single-stage microbiological sampler with tryptic soy agar (Difco Laboratories, Detroit, MI, USA) and malt extract agar (Difco Laboratories, Detroit, MI, USA).
  Airborne endotoxin and mite samples were collected using 1-µm pore polytetrafluoroethylene (Teflon) membrane filters (Pall Corporation, Port Washington, NY, USA) placed in disposable plastic cassettes (37 mm; HIBLOW SPP-25 GA, Techno Takatsuki, Japan).
Fractional exhaled nitric oxide (FeNO) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  FeNO, considered an indicator of airway inflammation, was measured using the NIOX VERO device (Aerocrine AB, Solna, Sweden).
Blood pressure | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We employed the HEM-8712 device (Omron Healthcare Co. Ltd., Japan) to measure blood pressure.
Heavy metals | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We assessed 15 heavy metals in urine samples, including Cr, Mn, Fe, Co, Ni, As, Se, Rb, Sr, Cd, Cs, V, Cu, Zn, Mo, using an inductively coupled plasma mass spectrometer (ICP-MS, X-series II, Thermo Fisher Scientific, Germany).
Polycyclic aromatic hydrocarbons | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We used SCIEX 4000QTRAP Triple Quadrupole Hybrid Linear Ion Trap Mass Spectrometer to assess urinary polycyclic aromatic hydrocarbons, including 1-hydroxypyrene, 2-Hydroxyfluorene, 1-Hydroxyphenanthrene, 4-Hydroxyphenanthrene.
microRNA | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We evaluated miRNA, such as miR-146a-5p, miR-199a-5p, miR-21-5p, miR-222-3p, miR-155-5p, miR-29b-3p, miR-194-3p, using real time quantitative polymerase chain reaction (StepOnePlus™ Real-Time PCR System).
cell-free DNA | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We evaluated cell-free DNA, using real time quantitative polymerase chain reaction (StepOnePlus™ Real-Time PCR System).
Cytokines | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  We evaluated cytokines, including IL-6, IL-8, IL-10, IL-13, IL-17A, IL-17F, IL-22, IL-25, IL-28A, IL-29, IL-31, IL-33, IL-34, and TGF-β1, using (Enzyme-linked immunosorbent assay, ELISA) assay (R & D Systems, Minneapolis, MN).
slow vital capacity (SVC) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
forced expiratory volume in 1 s (FEV1) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed.
forced vital capacity (FVC) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed.
FEV1/FVC | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
peak expiratory flow (PEF) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
maximal mid-expiratory flow (MMEF) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
forced expiratory flow (FEF) at 25% (FEF25) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
FEF50 | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
FEF75 | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  A multifunction spirometer (HI-801, Chest MI, Tokyo, Japan) was employed to assess the lung function.
asthma control test (ACT) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  The asthma control test (ACT) served as a measure of asthma control, with high scores indicating better control of the condition.
Respiratory symptoms score | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  The respiratory symptoms score evaluated in the questionnaire were stuffy nose, sneezing, runny nose, cough, shortness of breath, and chest tightness. The participants were asked to rate the severity of each respiratory symptom by using a 4-point scale, where 0, 1, 2, and 3 denoted no, mild, moderate, and severe symptoms, respectively.
COPD Assessment Test (CAT) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  The COPD Assessment Test (CAT) includes eight items (cough, sputum, breathlessness, chest tightness, confidence, activity, sleep and energy levels), rated on a 5-point scale (1 to 5).
modified Medical Research Council Dyspnea Scale (mMRC) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  The modified Medical Research Council Dyspnea Scale (mMRC) assessed dyspnea using a 5-grade scale (Grade 0 to Grade 4).
Breathlessness, Cough, and Sputum Scale (BCSS) | On day 0 ( before intervention), day 7 and day 13 ( after intervention)
  The Breathlessness, Cough, and Sputum Scale (BCSS) evaluated cough, sputum, and breathlessness using a 5-point scale (0 to 4).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not publicly available due to privacy and ethical restrictions.